CLINICAL TRIAL: NCT04432597
Title: Phase I/II Trial of HPV Vaccine PRGN-2009 Alone or in Combination With Anti-PD-L1/TGF-Beta Trap (M7824) in Subjects With HPV Positive Cancers
Brief Title: HPV Vaccine PRGN-2009 Alone or in Combination With Anti-PDL1/TGF-Beta Trap (M7824) in Subjects With HPV Associated Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Charalampos Floudas, MD, DMSc, MS, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200104; 20-C-0104
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: HPV Positive Cancer; Vulvar, Vaginal, Penile, Rectal Cancer; Anal Cancer; Oropharyngeal Cancer; Cervical Cancer
Keywords: HPV Associated Malignancy; Immunotherapy; HPV Vaccine; PRGN-2009; M7824
MeSH Terms: conditions — Rectal Neoplasms; Anus Neoplasms; Oropharyngeal Neoplasms; Uterine Cervical Neoplasms | interventions — Electrocardiography; Biopsy; Tomography, X-Ray Computed; Magnetic Resonance Imaging; Dexamethasone; Calcium Dobesilate; Epinephrine; Diphenhydramine; Ibuprofen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1/Arm 1A (Experimental): Human Papillomavirus Vaccine (HPV) vaccine at 1x10(11) Viral Particles (VP) Dose Level 1 (DL1) and at 5x10(11) VP Dose Level 2 (DL2)
  Interventions: Biological: PRGN-2009; Diagnostic Test: EKG; Procedure: Biopsy; Diagnostic Test: CT Scan; Diagnostic Test: MRI; Drug: Brain CT; Drug: Brain MRI; Drug: Dexamethasone; Drug: Epinephrine; Drug: Diphenhydramine; Drug: Ibuprofen
- 2/Arm 1B (Experimental): Human Papillomavirus Vaccine (HPV) vaccine at recommended phase 2 dose (RP2D) plus M7824 at 1200 mg.
  Interventions: Biological: PRGN-2009; Biological: M7824; Diagnostic Test: EKG; Procedure: Biopsy; Diagnostic Test: CT Scan; Diagnostic Test: MRI; Drug: Brain CT; Drug: Brain MRI; Drug: Dexamethasone; Drug: Epinephrine; Drug: Diphenhydramine; Drug: Ibuprofen
- 3/Arm 2A (Experimental): Human Papillomavirus Vaccine (HPV) vaccine at recommended phase 2 dose (RP2D) given as neoadjuvant or induction therapy.
  Interventions: Biological: PRGN-2009; Diagnostic Test: EKG; Procedure: Biopsy; Diagnostic Test: CT Scan; Diagnostic Test: MRI; Drug: Brain CT; Drug: Brain MRI; Drug: Dexamethasone; Drug: Epinephrine; Drug: Diphenhydramine; Drug: Ibuprofen
- 4/Arm 2B (Experimental): Human Papillomavirus Vaccine (HPV) vaccine at recommended phase 2 dose (RP2D) plus M7824 at 1200 mg given as neoadjuvant or induction therapy.
  Interventions: Biological: PRGN-2009; Biological: M7824; Diagnostic Test: EKG; Procedure: Biopsy; Diagnostic Test: CT Scan; Diagnostic Test: MRI; Drug: Brain CT; Drug: Brain MRI; Drug: Dexamethasone; Drug: Epinephrine; Drug: Diphenhydramine; Drug: Ibuprofen

INTERVENTIONS:
Biological: PRGN-2009 — On the phase I portion of the protocol PRGN-2009 will be administered on Day (D)1, D15, D29 followed by booster vaccines every 4 weeks for up to a year. The dose level given as booster will be the same dose participants will be receiving for D1, D15 and D29. On the phase II portion of the protocol PRGN-2009 will be administered on just D1 and D15 for Cohort 1/Arm 1A, Cohort 2/Arm 1B, Cohort 3/Arm 2A, and Cohort 4/Arm2B.
Biological: M7824 — Subjects enrolled to Cohort 2/Arm 1B will receive M7824 (MSB0011359C) via intravenous (IV) infusion over 1 hour (-10 minutes / +20 minutes, that is, over 50 to 80 minutes) once every 2 weeks. M7824 will be administered as a "flat" dose of 1,200 mg independent of body weight. M7824 is administered as an intravenous infusion with a mandatory 0.2 micron in-line filter.
  Other Names: MSB0011359C
  Arms: 2/Arm 1B; 4/Arm 2B
Diagnostic Test: EKG — Screening, end of treatment and follow-up.
  Other Names: Electrocardiogram
Procedure: Biopsy — For immune analysis: Baseline Day 1 and odd numbered weeks (week(W) 1, W3, W5, W7 onwards.
  Other Names: Bx
Diagnostic Test: CT Scan — CT scan chest, abdomen, pelvis, neck, and/or skull as clinically indicated. Tumor evaluation at screening, baseline Day 1, odd numbered weeks (week(W) 1, W3, W5, W7 onwards. Long term follow-up.
  Other Names: Computed tomography
Diagnostic Test: MRI — Tumor evaluation at screening, baseline Day 1, odd numbered weeks (week(W) 1, W3, W5, W7 onwards. Long term follow-up.
  Other Names: Magnetic resonance imaging
Drug: Brain CT — Screening. As clinically indicated in participants with known central nervous system (CNS) disease.
  Other Names: Brain computed tomography
Drug: Brain MRI — Screening. As clinically indicated in participants with known central nervous system (CNS) disease.
  Other Names: Brain magnetic resonance imaging
Drug: Dexamethasone — Dexamethasone 10mg for hypersensitivity reactions.
  Other Names: Decadron; Ozurdex; Dexycu
Drug: Epinephrine — 1:1,000 dilution for hypersensitivity reactions.
  Other Names: Adrenaline
Drug: Diphenhydramine — Antihistamines (e.g., Diphenhydramine) given intravenously for allergy.
  Other Names: Benadryl
Drug: Ibuprofen — For flu-like symptoms. 400mg or comparable Nonsteroidal anti-inflammatory drugs (NSAID) dose, may be administered 2 hours before and 8 hours after the start of each intravenous infusion.
  Other Names: Advil; Motrin IB; Midol IB

SUMMARY:
Background:

For some cancers associated with human papillomavirus (HPV), standard treatments are not helpful. Researchers want to see if a vaccine for HPV combined with a drug called M7824 (MSB0011359C) has a better effect on these cancers than when they work alone.

Objective:

To find a safe dose of HPV vaccine alone or combined with M7824. Also, to test if either HPV vaccine alone or combined with M7824 causes a better immune response.

Eligibility:

People ages 18 and older with locally advanced or metastatic HPV associated cancer (Phase I) or stage II or III p16-positive oropharyngeal cancer (Phase II)

Design:

Participants will be screened with:

Medical history

Physical exam

Blood, urine, and heart tests

Possible photos of skin lesions

Computed tomography (CT), magnetic resonance imaging (MRI), or nuclear bone scan: Participants will lie in a machine that takes pictures of the body. For the CT scan, they may have a contrast agent injected into a vein.

Participants may have up to 2 tumor biopsies. For participants in Phase II, this may be performed with a thin tube placed through the nose into the airway.

Participants will receive the HPV vaccine alone or with M7824. For participants on the Phase II, they will receive two doses of HPV vaccine under the skin either alone or with M7824 as an infusion spaced two weeks apart. This will be done prior to their planned chemoradiation or surgery. For participants on the Phase I, they will get the HPV vaccine injected under the skin 2 to 3 times in the first month. Then they will have a booster every 4 weeks. They will receive M7824 as an infusion into a vein every 2 weeks. Treatment will last up to 1 year.

After they stop treatment, participants will have a visit within 4 weeks. They will then be contacted for long-term follow-up every year, for the rest of their lives.

...

DETAILED DESCRIPTION:
Background

* Metastatic human papillomavirus (HPV) associated malignancies (cervical, anal, oropharyngeal cancers, etc.) are often incurable and poorly palliated by standard therapies.
* HPV-positive (p16+) oropharyngeal cancers are the most common HPV-associated malignancy in the United States and are increasing in incidence.
* Stage II and III HPV-positive oropharyngeal cancer is primarily treated with definitive therapy.
* Although the prognosis for stage I HPV+ oropharyngeal cancer is favorable, about 20 percent of patients with stage II disease and 35 percent of patients with stage III disease will die within four years.
* Attempts to de-intensify treatment of HPV-positive oropharyngeal cancer by replacing high-dose cisplatin with cetuximab concurrent with radiotherapy have failed.
* Induction and neoadjuvant immunotherapy are an area of active study in this type of cancer. The aims of induction immunotherapy are to induce antigen-specific immunity prior to definitive therapy and to reduce the risk of disease relapse for patients with stage II and III disease.
* Therapeutic vaccines targeting HPV alone or in combination with M7824 (MSB0011359C) (dual programmed death-ligand 1 (PD-L1) and transforming growth factor beta (TGF- beta) inhibitor) have demonstrated induction of HPV antigen-specific responses and tumor growth inhibition in multiple pre-clinical models of HPV-positive malignancy.
* In clinical studies done in the Center for Cancer Research (CCR), M7824 as monotherapy has produced a notable objective response rate (35-40%) for metastatic HPV + cancers including Oropharyngeal Squamous Cell Carcinoma (OPSCC) and preclinical studies support the addition of an investigational HPV vaccine with therapeutic intent (PRGN-2009, a gorilla adenoviral based vaccine) to further increase anti-tumor efficacy.

Objectives:

Phase I in participants with recurrent/metastatic HPV positive cancer:

-Primary objective: To determine the safety and recommended phase II dose (RP2D) of PRGN-2009 (HPV vaccine) alone or in combination with M7824 administered at RP2D of 1200 mg every 2 weeks (q2w).

Phase II in participants with newly diagnosed stage I (T1, T2 N1)/II/III p16-positive oropharyngeal cancer and patients with newly diagnosed operable stage II/III/IVA/IVB/HPV + sinonasal squamous cell cancer:

-Primary objective: To determine if HPV vaccine alone (Arm 2A) is able to result in a >= 2-fold increase in cluster of differentiation 3 (CD3+) tumor infiltrating T cells post treatment compared with pre-treatment in p16-positive oropharyngeal cancer.

Eligibility:

Phase I:

* Men or women of age >= 18 years old.
* Subjects with cytologically or histologically confirmed locally advanced not amenable to potentially curative local therapies or metastatic HPV associated malignancies:

  * Cervical cancers;
  * p16+ Oropharyngeal cancers;
  * Anal cancers;
  * Vulvar, vaginal, penile, and squamous cell rectal cancers
  * Other locally advanced or metastatic solid tumors (e.g., lung, esophagus) that are known HPV+.
* Prior first line systemic therapy is required

Phase II:

* Men or women of age >= 18 years old.
* Subjects with newly diagnosed stage I (T1, T2 N1), II or III, II or III p16-positive oropharyngeal squamous cell carcinoma (OPSCC) or stage II/III/IVA/IVB HPV-SNSCC planned for definitive therapy.

Design:

Phase I: Recurrent/metastatic HPV associated cancer:

* A 3+3 dose escalation design will be used which will evaluate PRGN-2009 (HPV vaccine) at two dose levels (1x10^11 and 5x10^11 viral particle (VP) units) given as monotherapy followed by a third dose level evaluating the RP2D dose of PRGN-2009 in combination with 1200 mg (RP2D) of M7824. In addition, the combination of PRGN-2009 at RP2D with 1200 mg of M7824 will be expanded to a total of 10 evaluable participants to gauge the preliminary efficacy of the combination of PRGN-2009 and M7824 in participants with advanced disease.
* There will be a 4-week dose limiting toxicity (DLT) evaluation period for each dose level.
* It is expected that up to 22 participants may enroll.

Phase II:

Newly diagnosed p16-positive oropharyngeal cancer:

* Evaluation of HPV vaccine alone (Arm 2A: Stage I (T1,T2 N1)/II/III) as neoadjuvant/ induction therapy before definitive standard of care therapy.
* Participants will receive neoadjuvant/ induction immunotherapy at National Institutes of Health (NIH) Clinical Center and then be referred back to their home institution for definitive standard of care therapy.
* It is expected that up to 20 participants may enroll.
* Newly diagnosed stage II/III/IVA/IVB HPV-SNSCC:
* Enrollment and treatment will occur similarly as participants with p16+oropharyngeal cancer for exploratory correlates to advise possible future trials. Up to 2 participants may enroll in this group.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects with cytologically or histologically confirmed locally advanced not amenable to potentially curative local therapies or metastatic human papillomavirus (HPV) associated malignancies (Phase I only):

  * Cervical cancers;
  * p16+ Oropharyngeal cancers;
  * Anal cancers;
  * Vulvar, vaginal, penile, and squamous cell rectal cancers;
  * Other locally advanced or metastatic solid tumors (e.g., lung, esophagus) that are known HPV+.
* Subjects with cytologically or histologically confirmed newly diagnosed stage II or III p16-positive oropharyngeal squamous cell carcinoma planned for definitive therapy or with newly diagnosed stage II or III or IVA or IVB HPV-positive sinonasal squamous carcinoma (HPV-SNSCC) eligible for primary surgery (Phase II only).
* Subjects must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Phase 1 only).
* Phase I only: Participants must have received one prior line of systemic chemotherapy in the recurrent/metastatic setting as well as checkpoint blockade therapy in tumors with Food and Drug Administration (FDA) approval (head and neck squamous cell cancer and programmed death-ligand 1 (PDL1+) cervical cancer). Exceptions to this include participants not eligible to receive standard therapy.
* Men or Women; Age >=18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Adequate hematologic function at screening, as follows:

  * Absolute neutrophil count (ANC) >=1 x 109/L;
  * Hemoglobin >= 9 g/dL;
  * Platelets >= 75,000/microliter.
* Adequate renal and hepatic function at screening, as follows:

  * Serum creatinine =< 1.5 x upper limit of normal (ULN) OR Measured or calculated creatinine clearance >= 40 mL/min for participant with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl);
  * Bilirubin =< 1.5 x ULN OR in subjects with Gilbert's syndrome, a total bilirubin =< 3.0 x ULN;
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN, unless liver metastases are present, then values must be =< 3 x ULN).
* The effects of the immunotherapies (PRGN-2009 vaccine and M7824) on the developing human fetus are unknown. For this reason and because M7824 and PRGN-2009 used in this trial are possibly teratogenic, women of child-bearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and up to 2 months following the last dose of M7824 study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participants serologically positive for human immunodeficiency virus (HIV), Hep B, Hep C are eligible as long as the viral loads are undetectable by quantitative polymerase chain reaction (PCR). HIV positive participants must have cluster of differentiation 4 (CD4) count >= 200 cells per cubic millimeter at enrollment, be on stable antiretroviral therapy for at least 4 weeks and have no reported opportunistic infections or Castleman's disease within 12 months prior to enrollment.

EXCLUSION CRITERIA:

* Participants with prior investigational drug, live vaccine, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 28 days prior to the first drug administration except if the investigator has assessed that all residual treatment-related toxicities have resolved or are minimal and feel the participant is otherwise suitable for enrollment. Participants may continue adjuvant hormonal therapy in the setting of a definitively treated cancer (e.g., breast).
* Major surgery within 28 days prior to the first drug administration (minimally invasive procedures such as diagnostic biopsies are permitted).
* Known active brain or central nervous system metastasis (less than a month out from definitive radiotherapy or surgery), seizures requiring anticonvulsant treatment (<3 months) or clinically significant cerebrovascular accident (<3 months). In order to be eligible participants must have repeated central nervous system (CNS) imaging at least a month after definitive treatment showing stable CNS disease. Participants with evidence of intra-tumoral or peritumoral hemorrhage on baseline imaging are also excluded unless the hemorrhage is grade =< 1 and has been shown to be stable on two consecutive imaging scans.
* Pregnant women are excluded from this study because M7824 and PRGN-2009 vaccine have not been tested in pregnant women and there is potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these immunotherapies, breastfeeding should be discontinued if the mother is treated on this protocol.
* Only for Phase I, Arm 1B: Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with exception of:

  * Diabetes type I, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease or other mild autoimmune disorders not requiring immunosuppressive treatment;
  * Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable;
  * Subjects on systemic intravenous or oral corticosteroid therapy with the exception of

physiologic doses of corticosteroids (=< the equivalent of prednisone 10 mg/day) or other immunosuppressors such as azathioprine or cyclosporin A are excluded on the basis of potential immune suppression. For these subjects these excluded treatments must be discontinued at least 1 weeks prior to enrollment for recent short course use (=< 14 days) or discontinued at least 4 weeks prior to enrollment for long term use (> 14 days). In addition, the use of corticosteroids as premedication for contrast-enhanced studies is allowed prior to enrollment and on study.

* Only for Phase I: Subjects with a history of serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, bleeding diathesis or recent (within 3 months) clinically significant bleeding events, known left ventricular ejection fraction <50% (confirmation of ejection fraction (EF) > 50% is not required for eligibility), history of myocarditis, or recent myocardial infarction (within 6 months), or other illness considered by the Investigator as high risk for M7824 drug treatment.
* Only for Phase I: Subjects refusing to accept blood products as medically indicated.
* History of second malignancy within 3 years of enrollment except for the following: adequately treated localized skin cancer, cervical carcinoma in situ, superficial bladder cancer, other localized malignancy which has been adequately treated or malignancy which does not require active systemic treatment (e.g., low risk chronic lymphocytic leukemia (CLL)). For participants enrolled on the phase I portion of the protocol a second HPV driven malignancy is allowed.
* Only for Phase I, Arm 1B: Subjects with a known severe hypersensitivity reaction to monoclonal antibodies or its excipients (grade >/= 3 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v5) will be evaluated by the allergy/immunology team prior to enrollment.
* Prior allogenic tissue/solid organ transplant.
* For participants who may receive M7824: previous life-threatening side effects resulting from prior checkpoint inhibitor therapy.
* Participants with pulse oximetry < 92% on room air at screening.
* Participants unable to provide informed consent.
* Participants whose inclusion in the trial would in the judgement of the principal investigator (PI) lead to time from diagnosis to initiation of curative treatment of>70 days (Arm 2A only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety and recommended phase II dose of PRGN-2009 | one year
  Phase I: In participants with recurrent/metastatic HPV positive cancer - To determine the safety and recommended phase II dose (RP2D) of PRGN-2009 (HPV vaccine) alone or in combination with M7824 administered at RP2D of 1200 mg q2w.
Level increase in CD3+ tumor infiltrating T cells post-treatment compared to pre-treatment | one year
  Phase II: In participants with newly diagnosed stage I (T1,T2 N1)/II/III p16-positive oropharyngeal cancer - To determine if HPV vaccine alone (Arm 2A) is able to result in a equal to or greater than 2-fold increase in CD3+ tumor infiltrating T cells post treatment compared with pre-treatment in p16-positive oropharyngeal cancer.

SECONDARY OUTCOMES:
ratio of participants that are hospitalized because of adverse events attributed to disease progression | study end
  Phase 1: To assess ratio of participants that are hospitalized because of adverse events attributed to disease progression.
3-year overall and relapse-free survival rate for PRGN-2009 alone | study end
  Phase II: To determine the 3-year overall and relapse-free survival rate for PRGN-2009 alone (Arm 2A) as neoadjuvant/ induction therapy before definitive standard of care therapy for this population.
overall survival (OS) | study end
  Phase 1: To assess overall survival (OS).
progression-free survival time (PFS) | study end
  Phase 1: To assess progression-free survival time (PFS).
duration of response | study end
  Phase 1: To assess duration of response.
assess the safety of the recommended phase II dose (RP2D) of PRGN-2009 (HPV vaccine) alone | study end
  Phase II: To assess the safety of the recommended phase II dose (RP2D) of PRGN-2009 (HPV vaccine) alone in this participant population.
does the use of PRGN-2009 alone result in significantly prolonged survival | study end
  Phase II: To determine if the use of PRGN-2009 alone results in significantly prolonged survival as compared to the expected 80% three-year historical survival for this population.
overall response rate (ORR) | study end
  Phase 1: To assess overall response rate (ORR) according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Floudas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Floudas CS, Goswami M, Donahue RN, Strauss J, Pastor DM, Redman JM, Brownell I, Turkbey EB, Steinberg SM, Cordes LM, Marte JL, Khan MH, McMahon S, Lamping E, Manu M, Manukyan M, Brough DE, Lankford A, Jochems C, Schlom J, Gulley JL. PRGN-2009 and bintrafusp alfa for patients with advanced or metastatic human papillomavirus-associated cancer. Cancer Immunol Immunother. 2025 Mar 21;74(5):155. doi: 10.1007/s00262-025-04009-z. PMID 40116923
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0104.html

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT04432597/Prot_SAP_003.pdf
  • Informed Consent Form: Phase I Participants Consent (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT04432597/ICF_001.pdf
  • Informed Consent Form: Phase II Participants Consent (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT04432597/ICF_002.pdf